CLINICAL TRIAL: NCT01306916
Title: Coexisting Thyroid Disease and Hyperparathyroidism
Status: Completed | Type: Observational
Sponsor: Walter Reed Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Alexander Stojadinovic, Director, Combat Wound Initiative Program, Walter Reed National Military Medical Center
Other Study IDs: 04-20018
Record Dates: First submitted 2011-01-12; First posted 2011-03-02 (Estimated); Last update posted 2012-07-03 (Estimated); Status verified 2012-07

CONDITIONS: Hyperthyroidism
Keywords: thyroid disease, hyperthyroidism
MeSH Terms: conditions — Hyperthyroidism; Thyroid Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1 of 1: diagnosis of primary and secondary hyperparathyroidism scheduled to undergo parathyroid resection.

SUMMARY:
Purpose: Prospective studies of patients with hyperparathyroidism are warranted to determine the prevalence of concurrent thyroid disease applying the current standard of pre-operative radioscintigraphic and sonographic imaging of the neck. Timely diagnosis and treatment of co-existing thyroid disease is advantageous given the well-established increased morbidity associated with a second neck exploration. The purpose of this study is to determine the prevalence and specific type of thyroid disease in patients with hyperparathyroidism, and to determine the frequency with which the presence of thyroid disease alters the treatment plan for patients with hyperparathyroidism.

Research Design: This will be a prospective single arm observational study of up to 200 military health care beneficiaries over the age of 18 years with primary and secondary hyperparathyroidism scheduled to undergo parathyroid resection.

Methodology: Patients will undergo standard pre-operative imaging of the neck including ultrasonography and 99mTc-sestamibi scintigraphy. An operative plan will be developed based on the information obtained from history, physical examination, laboratory studies, and imaging studies. The number and type of thyroid disease in these patients will be determined based on these non-invasive studies (Objective A). A change in the otherwise standard treatment will include those patients having partial or complete resections of their thyroid glands because: a) the patients would have undergone minimally invasive surgery if not for the results of the imaging studies, and, b) the patients who would have undergone 3 ½ gland parathyroidectomy if not for the results of the imaging studies (Objective B).

ELIGIBILITY:
Inclusion Criteria:

Patients with hyperparathyroidism and appropriate indications for operation

* Patients over 18 years of age and capable of providing informed consent
* Each patient must provide written informed consent prior to entering the study.

Exclusion Criteria:

* Patients who have previously undergone thyroid or parathyroid operation
* Patients with medullary thyroid carcinoma and hyperparathyroidism or suspected multiple endocrine neoplasm syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 200 military health care beneficiaries over the age of 18 years with primary and secondary hyperparathyroidism scheduled to undergo parathyroid resection.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2004-09; Primary Completion 2010-12 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
To determine the prevalence and specific type of thyroid disease in patients with hyperparathyroidism. | One year

SECONDARY OUTCOMES:
To determine the frequency with which the presence of thyroid disease alters the treatment plan for patients with hyperparathyroidism. | One year

CONTACTS AND LOCATIONS:
Locations (1):
- Walter Reed Army Medical Center, Washington D.C., District of Columbia, United States